CLINICAL TRIAL: NCT07317297
Title: Extracorporeal Shockwave Therapy in the Treatment of Peyronie's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Doç.Dr.Ömer Şevgin, Assoc.Prof.Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar79
Record Dates: First submitted 2025-12-18; First posted 2026-01-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Peyronie Disease
MeSH Terms: conditions — Penile Induration | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): patients receiving normal routine pharmacological treatment without any special intervention
  Interventions: Other: control
- Extracorporeal Shockwave Therapy (Experimental): Patients receiving Extracorporeal Shockwave Therapy treatment
  Interventions: Other: Extracorporeal Shockwave Therapy

INTERVENTIONS:
Other: Extracorporeal Shockwave Therapy — Extracorporeal Shockwave Therapy will follow a standard protocol. The treatment is planned as a total of 8 sessions (3000 pulses per session, 2.5 bar pressure, 15 Hz frequency) twice a week using a radial shockwave device. Focusing will be done on the penile shaft via gel according to the plaque localization, and shock waves will be applied to the plaque area.
  Arms: Extracorporeal Shockwave Therapy
Other: control — patients receiving normal routine pharmacological treatment without any special intervention
  Arms: control

SUMMARY:
Investigation of the effectiveness of extracorporeal shock wave therapy in the treatment of Peyronie's disease.

DETAILED DESCRIPTION:
The study is designed as a single-center, prospective clinical trial. Participants will be selected from among patients who present to the clinic and are diagnosed with stable stage Peyronie's disease. All participants who meet the eligibility criteria and provide written consent will undergo a standard Extracorporeal Shockwave Therapy protocol. All participants will be evaluated before and after treatment using the International Erectile Function Index-5 and the Quality of Life Questionnaire short form. The results will be statistically analyzed and interpreted.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals aged 18-65 years.
* Having been diagnosed with Peyronie's Disease that has been stable (without increasing pain and curvature) for at least 6 months.
* Presence of palpable penile plaque.

Exclusion Criteria:

* Acute inflammatory stage (painful, progressive)
* Having previously undergone surgery, needle therapy (e.g., Xiaflex), or Extracorporeal Shockwave Therapy for peyronie's disease.
* Uncontrolled diabetes, severe coagulopathy, or receiving anticoagulant therapy.
* History of penile cancer.
* Severe erectile dysfunction.
* Patients who are considered unable to comply with the study protocol or who cannot attend follow-up visits.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — diseases specific to men
Enrollment: 50 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Erectile function | 5 weeks
  The International Index of Erectile Function is recorded as a total score. It is measured by a self-reported questionnaire with 5 domains, with each domain consisting of 5 options. The score ranges from 5 to 25, with 5 being the lowest score (severe erectile dysfunction) and 25 being the best score (maximal erection)
Short Form-36 | 5 weeks
  Short Form-36 Health Survey is a non-disease-specific instrument consisting of 36 items used to assess health-related quality of life. It includes eight subscales covering physical and mental health domains. Each subscale is scored from 0 to 100, with higher scores indicating better health status, while one item assessing health change is not included in subscale scoring. A high score indicates a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Azizov, Study Chair — Uskudar University
Locations (1):
- Koreya Serq Tebabeti, Baku, Azerbaijan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ergun M, Sagir S. Low-Intensity Extracorporeal Shock Wave Therapy and Platelet-Rich Plasma: Effective Combination Treatment of Chronic-Phase Peyronie's Disease. Arch Esp Urol. 2025 Mar;78(2):164-169. doi: 10.56434/j.arch.esp.urol.20257802.23. PMID 40191859
- [Background] Porst H. Review of the Current Status of Low Intensity Extracorporeal Shockwave Therapy (Li-ESWT) in Erectile Dysfunction (ED), Peyronie's Disease (PD), and Sexual Rehabilitation After Radical Prostatectomy With Special Focus on Technical Aspects of the Different Marketed ESWT Devices Including Personal Experiences in 350 Patients. Sex Med Rev. 2021 Jan;9(1):93-122. doi: 10.1016/j.sxmr.2020.01.006. Epub 2020 Jun 2. PMID 32499189
- [Background] Rosenberg JE, Ergun O, Hwang EC, Risk MC, Jung JH, Edwards ME, Blair Y, Dahm P. Non-surgical therapies for Peyronie's disease. Cochrane Database Syst Rev. 2023 Jul 17;7(7):CD012206. doi: 10.1002/14651858.CD012206.pub2. PMID 37490423